CLINICAL TRIAL: NCT05841459
Title: Study of Spiritual Well-being, Self-compassion, Physical Symptoms Distress and Demoralization Among Hemodialysis Patients
Brief Title: Spiritual Well-being, Self-compassion, Physical Symptoms Distress and Demoralization Among HD Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ya-Chu Hsiao, professor, Chang Gung University of Science and Technology
Other Study IDs: 202212044RIND; NCT06097858 (obsolete NCT alias)
Record Dates: First submitted 2023-04-19; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Demoralization
Keywords: spirituality; self-compassion; demoralization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the associations between spiritual well-being, self-compassion, physical symptoms distress and demoralization among hemodialysis patients

DETAILED DESCRIPTION:
The aims of this study is to explore the associations between spiritual well-being, self-compassion, physical symptom distress and demoralization in hemodialysis patients.

A cross-sectional correlation design will be used. We use convenient sample to recruit hemodialysis patients in a regional teaching hospital in the southern Taiwan. The research data is collected with a pact of self-administrated questionnaire including Chinese version of the Demoralization Scale , FACITsp-12 Scale, Self-Compassion Scale, and Physical Symptom Distress Scale. SPSS statistical software will be used to data analysis. Analysis methods included descriptive and inferential statistics. Finally, multiple linear regression will be used to test the predictors of demoralization. The research results will offer health providers to identify symptoms related to demoralization earlier and provide appropriate care to patients to adapt the long treatment process and improve their quality of life

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patient who agrees to join this study.
* The participant is over 20 years old.
* The participant has a clear consciousness and can communicate in Mandarin and Taiwanese to answer the questionnaire.

Exclusion Criteria:

* The hearing impaired cannot communicate.
* Intensive care unit or inpatients.
* Mental disorders or dementia such as depression, schizophrenia, and anxiety diagnosed by a physician.
* Those who are seriously unwell or have unstable vital signs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
demoralization | during the procedure
  The demoralization scale is a validated multidimensional measure that assesses patients' status of demoralization

SECONDARY OUTCOMES:
spiritual well-being | during the procedure
  The spiritual well-being scale is a validated multidimensional measure that assesses patients' spirituality
self compassion | during the procedure
  The self-compassion scale is a validated multidimensional measure that assesses patients' level of self-compassion
physical symptom distress | during the procedure
  The physical symptom distress scale is a validated multidimensional measure that assesses patients' level of physical symptom distress

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Chu Hsiao, EdD, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan, N/A = Not Applicable, Taiwan

IPD SHARING:
Plan to Share IPD: No